CLINICAL TRIAL: NCT00412425
Title: Evaluation of Two Different Schedules of Palonosetron for the Prevention of Nausea and Vomiting in Patients With Metastatic Melanoma Receiving Concurrent Biochemotherapy
Brief Title: Palonosetron for Prevention of Biochemotherapy Induced Nausea and Vomiting
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0506
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Results first posted 2012-05-04 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-04

CONDITIONS: Melanoma
Keywords: Melanoma; Nausea; Vomiting; Palonosetron; Cisplatin; Vinblastine; Loss of Appetite; Weight loss
MeSH Terms: conditions — Melanoma; Nausea; Vomiting; Anorexia; Weight Loss | interventions — Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 Days Palonosetron (Active Comparator): 2 Days Palonosetron 0.25 mg intravenous (IV)
  Interventions: Drug: Palonosetron
- 3 Days Palonosetron (Active Comparator): 3 Days Palonosetron 0.25 mg IV
  Interventions: Drug: Palonosetron

INTERVENTIONS:
Drug: Palonosetron — 0.25 mg IV (By Vein) Daily for 2 Days or 0.25 mg IV Daily for 3 Days.

SUMMARY:
Primary Objectives:

* Safety of palonosetron administered for control of nausea and vomiting in patients with metastatic melanoma receiving biochemotherapy.
* To determine the patterns and severity of nausea and vomiting in two groups of patients with metastatic melanoma receiving biochemotherapy with palonosetron premedication using two schedules of palonosetron administration.

DETAILED DESCRIPTION:
Palonosetron is designed to work by blocking the substance serotonin from binding to the brain and gastrointestinal tract, which may help to decrease nausea and vomiting.

Participants in this study will be receiving biochemotherapy treatment as part of their routine care. This treatment will include 3 chemotherapy drugs (cisplatin, vinblastine, and DTIC) and 2 drugs that stimulate the immune system (interferon and interleukin-2 (IL-2)). Biochemotherapy often causes nausea, vomiting, loss of appetite, and weight loss. Palonosetron will be given on this study to try to treat the side effects of biochemotherapy.

If you agree to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of 2 treatment groups. You have an equal chance of being assigned to either group.

Participants in Group 1 will receive palonosetron by vein over a few minutes starting 30 minutes before receiving chemotherapy on Days 1 and 4 of therapy. Participants in Group 2 will receive palonosetron by vein over a few minutes on Days 1, 3, and 5.

All participants on this study will also receive Ativan by vein every 8 hours for 5 days. Ativan is given for additional control of nausea and it will also help to sedate you. In addition to palonosetron, you may be given standard anti-nausea medications such as lorazepam or compazine if you experience intolerable nausea and vomiting while on study.

You will also be asked to fill out a Functional Living Index-Emesis (FLIE) questionnaire every day for 7 days in a row. The questionnaire will ask about any nausea and/or vomiting you are experiencing and the effect of the therapy on your quality of life. You will stay in the hospital for at least 7 days while you receive treatment.

After the first course of palonosetron given with biochemotherapy, your doctor will decide if you will receive additional courses of palonosetron or if you will be given another anti-nausea drug.

If your doctor does decide to have you continue on palonosetron, it will be given off study. Your participation in this study will be over after 1 course.

This is an investigational study. Palonosetron has been approved by FDA for control of nausea and vomiting caused by chemotherapy. However, it has not been adequately evaluated for safety and effectiveness in patients receiving high dose interleukin-2 alone or in combination with chemotherapy. About 30 patients will take part in this study. All patients will enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* They have non-resectable stage III or IV metastatic melanoma with measurable disease and have agreed to be treated with biochemotherapy.
* They have Zubrod performance status of 0-1
* They have normal blood counts with a white blood count (WBC) count >/= 3,500/mm^3, ANC >/= 1,500/mm^3 and a platelet count >/= 100,000/mm^3 and have serum creatinine <1.5 mg/dl, and serum bilirubin level < 1.5 mg/dl, and no evidence of significant cardiac or pulmonary dysfunction.
* They have no significant intercurrent illness such as a serious infection, significant psychiatric illness, hypercalcemia (calcium >11 mg), gastro-intestinal (GI) bleeding or evidence of brain metastasis.
* They have not been exposed to prior interferon, interleukin-2 or previous chemotherapy including regional perfusion. Prior radiation therapy for metastatic melanoma is permitted provided the patient has unirradiated metastatic sites for response evaluation and has fully recovered from its toxicity.
* They must have been off corticosteroids for at least 2 weeks.

Exclusion Criteria:

* They are younger than 18 years or more than 65 years of age and those with an expected survival of less than 8 weeks or a Zubrod performance status of 2, 3 or 4.
* They have received previous treatment with any prior systemic chemotherapy for unresectable metastasis including and not limited to the following drugs: cisplatin, vinblastine, Dacarbazine (DTIC), interferon and interleukin-2
* They have active central nervous system involvement by melanoma either as brain metastasis, spinal cord compression, or meningeal carcinomatosis".
* They have significant cardiac illness such as symptomatic coronary artery disease or previous history of myocardial infarction, impaired left ventricular function or serious cardiac arrhythmias requiring therapy.
* They have significant impairment of pulmonary function on account of chronic bronchitis or chronic obstructive pulmonary disease (COPD).
* They have symptomatic effusions on account of pleural, pericardial or peritoneal metastasis of melanoma.
* They have history of a second malignant tumor (except for other skin cancers and in situ carcinoma of the cervix) within the past 5 years and uncertainty about the histologic nature of the metastatic lesions.
* They are on corticosteroids or any other type of immunosuppressive agent (e.g., methotrexate, chloroquine, azathioprine, cyclophosphamide).
* They are pregnant or breast feeding. Patients of childbearing potential must agree to use an effective method of contraception.
* They have known hypersensitivity to any of the study drugs or to other selective 5-HT3(subscript).
* They have ongoing emesis due to any organic etiology including but not limited to central nervous system or gastrointestinal metastasis.
* They have grade 2 or higher nausea due to administration of drugs including but not limited to narcotics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agop Y. Bedikian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 11/17/2006 - 8/1/2008. All recruitment done at UT MD Anderson Cancer Center.
Groups:
- 3 Days Palonosetron: 3 Days Palonosetron 0.25 mg intravenous (IV)
- 2 Days Palonosetron: 2 Days Palonosetron 0.25 mg IV
Period: Overall Study
Arm/Group | 3 Days Palonosetron | 2 Days Palonosetron
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 Days Palonosetron | 2 Days Palonosetron | Total
Number analyzed (Participants) | 15 | 15 | 30
Age Continuous [Median (Full Range); unit: years] | 55 [23 to 64] | 49 [33 to 65] | 53 [23 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 7 | 11 | 18
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Participants Response to Palonosetron
Description: Participants response measured as incidences biochemotherapy emesis and those of nausea interfering with appetite, sleep, physical activity, social life and enjoyment of life are summarized. Response evaluated during 5-day administration of biochemotherapy and the 23 subsequent days after therapy ends.
Time Frame: 7 days
Population: Analysis was per protocol.
Measure: Number; unit: episodes of nausea/vomiting
Arm/Group | 3 Days Palonosetron | 2 Days Palonosetron
Number analyzed (Participants) | 15 | 15
episodes of nausea/vomiting
  Nausea Episodes (First 7 days) | 85 | 139
  Vomiting Episodes (First 7 days) | 44 | 72

ADVERSE EVENTS:
Time Frame: 19 months
Arm/Group | 3 Days Palonosetron | 2 Days Palonosetron
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 15/15 | 14/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 Days Palonosetron (N=15) | 2 Days Palonosetron (N=15)
Nausea (Gastrointestinal disorders) | 15 (128) | 14 (207)
Vomiting (Gastrointestinal disorders) | 11 (57) | 13 (89)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No